CLINICAL TRIAL: NCT00967057
Title: ALLR3: An International Collaborative Trial for Relapsed and Refractory Acute Lymphoblastic Leukaemia (ALL)
Brief Title: Combination Chemotherapy in Treating Young Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CCLG-ALLR3; CDR0000642221 (Registry Identifier: PDQ (Physician Data Query)); ISCRTN45724312 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register)); EUDRACT-2004-000052-16; EU-20938
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-01

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Dexamethasone; Idarubicin; Methotrexate; Mitoxantrone; pegaspargase; Vincristine

ARMS (2):
- Arm I (induction therapy) (Experimental): Patients receive idarubicin IV over 1 hour on days 1 and 2; oral dexamethasone twice daily on days 1-5 and 15-19; intrathecal (IT) methotrexate on days 1 and 8; vincristine sulfate IV on days 3, 10, 17, and 24; and pegaspargase intramuscularly (IM) on days 3 and 17 or asparaginase IM on days 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25.
  Interventions: Drug: asparaginase; Drug: dexamethasone; Drug: idarubicin; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- Arm II (induction therapy) (Experimental): Patients receive mitoxantrone IV over 1 hour on days 1 and 2. Patients also receive dexamethasone, methotrexate, vincristine sulfate, and pegaspargase or asparaginase as in arm I.
  Interventions: Drug: asparaginase; Drug: dexamethasone; Drug: methotrexate; Drug: mitoxantrone hydrochloride; Drug: pegaspargase; Drug: vincristine sulfate

INTERVENTIONS:
Drug: asparaginase — Given intramuscularly
Drug: dexamethasone — Given orally
Drug: idarubicin — Given IV
  Arms: Arm I (induction therapy)
Drug: methotrexate — Given intrathecally
Drug: mitoxantrone hydrochloride — Given IV
  Arms: Arm II (induction therapy)
Drug: pegaspargase — Given intramuscularly
Drug: vincristine sulfate — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known which combination chemotherapy regimen is more effective in treating young patients with acute lymphoblastic leukemia.

PURPOSE: This partially randomized phase III trial is studying how well combination chemotherapy works in treating young patients with relapsed or refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the progression-free survival (defined as the time from study entry to the first occurrence of progression, relapse, death while in complete clinical remission, or second malignancy) of United Kingdom patients with relapsed or refractory acute lymphoblastic leukemia stratified by risk group.
* Evaluate whether a minimal residual disease (MRD) level of 10^-4 is a suitable criterion at the end of induction therapy on which to decide whether chemotherapy or stem cell transplantation will be most beneficial to patients with intermediate-risk disease.

Secondary

* Use MRD as a surrogate marker for response to therapy.

OUTLINE: This is a multicenter study. Patients are stratified by risk group (standard vs intermediate vs high) and participating country (UK and Ireland vs Australia and New Zealand vs The Netherlands).

Patients with standard-risk disease receive induction therapy, consolidation therapy, intensification therapy, interim maintenance therapy, and maintenance therapy. Patients with intermediate-risk disease receive induction therapy followed by assessment of minimal residual disease (MRD). Those whose MRD status is < 10^-4 at week 5 (after induction therapy) proceed to consolidation therapy followed by intensification therapy, interim maintenance therapy, and maintenance therapy. Those whose MRD status is ≥ 10^-4 at week 5 (after induction therapy) proceed to consolidation therapy followed by intensification therapy and assessment of MRD at week 13 (after intensification therapy). Those whose MRD status is ≥ 10^-3 at week 13 proceed to pre-stem cell transplantation cytoreduction (FLAD) followed by allogeneic stem cell transplant (ASCT). Those whose MRD status is < 10^-3 at week 13 proceed directly to ASCT. Patients with high-risk disease receive induction therapy, consolidation therapy, and intensification therapy followed by assessment of MRD at week 13 (after intensification therapy). These patients then proceed to further treatment (FLAD and/or ASCT) based on the same MRD parameters at week 13 as for patients with intermediate-risk disease.

* Induction therapy (weeks 1-4): Patients are randomized to 1 of 2 induction therapy arms.

  * Arm I: Patients receive idarubicin IV over 1 hour on days 1 and 2; oral dexamethasone twice daily on days 1-5 and 15-19; intrathecal (IT) methotrexate on days 1 and 8; vincristine sulfate IV on days 3, 10, 17, and 24; and pegaspargase intramuscularly (IM) on days 3 and 17 or asparaginase IM on days 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25.
  * Arm II: Patients receive mitoxantrone IV over 1 hour on days 1 and 2. Patients also receive dexamethasone, methotrexate, vincristine sulfate, and pegaspargase or asparaginase as in arm I.
* Consolidation therapy (weeks 5-8): Patients receive oral dexamethasone twice daily on days 1-5; vincristine sulfate IV on day 3; IT methotrexate on day 8; methotrexate IV continuously over 36 hours beginning on day 8; pegaspargase IM on day 9 or asparaginase IM on days 9, 11, 13, 15, 17, and 19; leucovorin calcium IV twice on day 10; and cyclophosphamide IV over 30 minutes and etoposide phosphate IV over 4 hours on days 15-19.
* Intensification therapy (weeks 9-13): Patients receive oral dexamethasone twice daily on days 1-5; vincristine sulfate IV on 3; IT methotrexate on days 1 and 22; cytarabine IV over 3 hours twice on days 1, 2, 8, and 9; asparaginase IM on days 2, 4, 9, 11, and 23; methotrexate IV continuously over 36 hours beginning on day 22; and leucovorin calcium IV twice on day 24.
* Interim maintenance therapy (weeks 14-29): Patients receive oral dexamethasone twice daily on days 1-5; IT methotrexate* on days 1 and 43; vincristine sulfate IV on day 3; high-dose oral methotrexate 4 times on day 22; oral leucovorin calcium twice on day 24; oral mercaptopurine once daily on days 1-42; oral methotrexate on days 8, 15, 29, and 36; oral thioguanine on days 43-49; etoposide phosphate IV over 4 hours and cyclophosphamide IV over 30 minutes on days 43 and 50; and cytarabine IV or subcutaneously (SC) on days 44-47 and 51-54. Treatment repeats every 56 days (8 weeks) for 2 courses.

Patients undergoing cranial irradiation do so before starting interim maintenance therapy. Patients undergoing testicular irradiation do so concurrently with interim maintenance therapy.

NOTE: *Patients who undergo cranial irradiation do not receive IT methotrexate.

* Maintenance therapy (weeks 30-117): Patients receive IT methotrexate* on day 15; oral dexamethasone twice daily on days 1-5, 29-33, and 57-61; vincristine sulfate IV on days 1, 29, and 57; oral mercaptopurine once daily on days 1-84; and oral methotrexate on days 1, 8, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 84 days (12 weeks) for 7 courses. Patients then receive 4 additional weeks (course 8) of maintenance therapy without IT methotrexate.

NOTE: *Patients who undergo cranial irradiation do not receive IT methotrexate.

* Pre-stem cell transplantation cytoreduction (FLAD): Patients receive fludarabine phosphate IV over 30 minutes and cytarabine over 4 hours on days 1-5 and liposomal daunorubicin citrate IV over 2 hours on day 1. Patients also receive filgrastim IV or SC beginning on day 7 and continuing until blood counts recover.
* ASCT: Patients undergo ASCT (including conditioning and graft-vs-host disease [GVHD] prophylaxis) according to national transplant guidelines based on the type of donor.
* Post-transplant immunotherapy: Patients who undergo ASCT may receive incremental doses of donor lymphocytes by infusion until a response and/or GVHD has occurred.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL) meeting 1 of the following criteria:

  * In first relapse after treatment

    * Has not yet received chemotherapy or radiotherapy for the first relapse
  * Primary refractory disease
* No mature B-cell ALL
* Meets criteria for one of the following risk groups:

  * Standard-risk disease: non-T-cell or T-cell ALL with late isolated extramedullary relapse
  * Intermediate-risk disease: non-T-cell ALL with early isolated extramedullary relapse or combined marrow and extramedullary relapse; non-T-cell ALL with late combined marrow and extramedullary relapse or isolated marrow relapse; or T-cell ALL with early isolated extramedullary relapse
  * High-risk disease: non-T-cell ALL with very early isolated extramedullary relapse, combined marrow and extramedullary relapse, or isolated marrow relapse; non-T-cell ALL with early isolated marrow relapse; T-cell ALL with very early isolated extramedullary relapse, combined marrow and extramedullary relapse, or isolated marrow relapse; T-cell ALL with early combined marrow and extramedullary relapse or isolated marrow relapse; or T-cell ALL with late combined marrow and extramedullary relapse or isolated marrow relapse

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bone marrow transplant

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 470 (Estimated)
Dates: Start 2002-10; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of United Kingdom (UK) patients stratified by risk groups
Evaluation of whether a minimal residual disease (MRD) level of 10(-4) is a suitable criterion at the end of induction therapy on which to decide whether chemotherapy or stem cell transplantation will be most beneficial to patients with intermediate- ...

SECONDARY OUTCOMES:
MRD as a surrogate marker for treatment response and PFS
Comparison of PFS, MRD level at day 35, and toxicity as response variables in patients randomized to receive induction therapy with mitoxantrone hydrochloride or idarubicin
PFS of all patients (UK, Dutch, Australian, and New Zealand) stratified by risk groups
Comparison of PFS and overall survival between patients enrolled in this study and patients enrolled in R2 or I-BFM
Evaluation of whether pre-stem cell transplantation cytoreduction (FLAD) reduces tumor load and how it affects outcome following transplant

CONTACTS AND LOCATIONS:
Overall Officials: Vaskar Saha, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (6):
- Women's and Children's Hospital, North Adelaide, South Australia, Australia
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Great Ormond Street Hospital for Children, London, England
  - Christie Hospital, Manchester, England
  - Southampton General Hospital, Southampton, England

REFERENCES:
- [Result] Parker C, Waters R, Leighton C, Hancock J, Sutton R, Moorman AV, Ancliff P, Morgan M, Masurekar A, Goulden N, Green N, Revesz T, Darbyshire P, Love S, Saha V. Effect of mitoxantrone on outcome of children with first relapse of acute lymphoblastic leukaemia (ALL R3): an open-label randomised trial. Lancet. 2010 Dec 11;376(9757):2009-17. doi: 10.1016/S0140-6736(10)62002-8. Epub 2010 Dec 3. PMID 21131038
- [Derived] Eckert C, Parker C, Moorman AV, Irving JA, Kirschner-Schwabe R, Groeneveld-Krentz S, Revesz T, Hoogerbrugge P, Hancock J, Sutton R, Henze G, Chen-Santel C, Attarbaschi A, Bourquin JP, Sramkova L, Zimmermann M, Krishnan S, von Stackelberg A, Saha V. Risk factors and outcomes in children with high-risk B-cell precursor and T-cell relapsed acute lymphoblastic leukaemia: combined analysis of ALLR3 and ALL-REZ BFM 2002 clinical trials. Eur J Cancer. 2021 Jul;151:175-189. doi: 10.1016/j.ejca.2021.03.034. Epub 2021 May 16. PMID 34010787
- [Derived] Parker C, Krishnan S, Hamadeh L, Irving JAE, Kuiper RP, Revesz T, Hoogerbrugge P, Hancock J, Sutton R, Moorman AV, Saha V. Outcomes of patients with childhood B-cell precursor acute lymphoblastic leukaemia with late bone marrow relapses: long-term follow-up of the ALLR3 open-label randomised trial. Lancet Haematol. 2019 Apr;6(4):e204-e216. doi: 10.1016/S2352-3026(19)30003-1. Epub 2019 Feb 27. PMID 30826273